CLINICAL TRIAL: NCT05497739
Title: Adjuvant Intraperitoneal Chemotherapy Guided by the Detection of Cancer Cell DNA in Peritoneal Lavage Fluid in Patients With Gastric Cancer: an Open-label, Phase 2 Trial
Brief Title: Intraperitoneal Chemotherapy Guided by the Detection of DNA in Peritoneal Lavage Fluid in Patients With Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong Bing Zhao, Senior doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/458-3129
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
Keywords: Peritoneal metastasis; Personalized mutation assay; Cancer cell DNA; Intraperitoneal Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal chemotherapy group (Experimental): In this study, patients with positive peritoneal lavage fluid cancer cell DNA will be given intraperitoneal chemotherapy followed by adjuvant systemic chemotherapy.
  Interventions: Drug: Intraperitoneal chemotherapy; Drug: Adjuvant systemic chemotherapy

INTERVENTIONS:
Drug: Intraperitoneal chemotherapy — 5-Fu 1 g/m^2 on Days 1, 8, 15, and 22; Albumin-paclitaxel 80-100 mg/time on Days 1, 8, 15, and 22; Cisplatin 25 mg/m^2 on Days 4, 11, 18, and 25; Interleukin-2 2 million units/time on Days 4, 11, 18, and 25.
Drug: Adjuvant systemic chemotherapy — Oxaliplatin 85 mg/m^2 on Day 1; S-1 depends on Body Surface Area (BSA), 40 mg Bid, Days 1-10 (BSA < 1.25 m^2), 50 mg Bid, Days 1-10 (BSA 1.25-1.50 m^2), 60 mg Bid, Days 1-10 (BSA > 1.50 m^2).

SUMMARY:
Peritoneal metastasis is a major pattern of gastric cancer recurrence and predicts poor prognosis. In our previous study, we developed a next-generation sequencing technology to detect minimal residual cancer cells in peritoneal lavage fluid with a personalized assay profiling tumor-specific mutations in patients with gastric cancer. With this technology, we predicted all the cases that developed peritoneal metastasis in patients with pT4 disease with 100% sensitivity and 91% specificity. Based on this result, a prospective phase 2 clinical trial is designed to evaluate the efficacy of adjuvant intraperitoneal chemotherapy in patients with positive cancer cell DNA detected in peritoneal lavage fluid by our personalized tumor-specific mutation profiling assay.

DETAILED DESCRIPTION:
Introduction:

Peritoneal metastasis is the most common pattern of gastric cancer recurrence and leads to rapid death. In a previous study, our team established a personalized method which could detect minimal cancer cell DNA in peritoneal lavage fluid with high sensitivity and specificity. We intend to perform a clinical trial to explore the efficacy of intraperitoneal chemotherapy on reducing the incidence of peritoneal metastases in patients with high risk defined by our personalized mutation detection method.

Methods and analysis:

This is a single-arm and single-center clinical trial. Sixty-eight patients with clinical T4 stage gastric cancers will be expected to be enrolled. During surgery, surgeons will wash upper abdominal cavity with 300-400 mL of normal saline before any manipulation of the tumor and collect about 200 mL peritoneal lavage fluid. Cancer cell DNA in peritoneal lavage fluid will be detected by next-generation sequencing using a personalized tumor-specific mutation profiling assay. Patients with positive peritoneal lavage fluid cancer cell DNA will receive adjuvant intraperitoneal chemotherapy in the second month since surgery, then followed by standard adjuvant systemic chemotherapy.

The primary endpoint is the incidence of peritoneal metastasis, and the secondary endpoints include peritoneal metastasis-free survival, disease-free survival (DFS), overall survival (OS), and the safety of intraperitoneal chemotherapy.

Ethics

This trial has been approved by the Ethics Committee of the National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College.

ELIGIBILITY:
Criteria:

1. Gastric adenocarcinoma confirmed by pathology (histology);
2. 18-75 years old;
3. Clinical T4 stage, no distant metastasis confirmed by CT and endoscopic ultrasonography (EUS), potentially curable by surgery;
4. Eastern Cooperative Oncology Group Performance Score 0 or 1;
5. Absolute neutrophil count at least 1.5×10^9/L; platelets count at least 80×10^9/L; hemoglobin at least 9 g/dL; serum creatinine or creatinine clearance no greater than 1.5 times upper normal limit (UNL); TSB no greater than 1.5 times ULN; AST (SGOT) and ALT (SGPT) no greater than 2.0 times ULN; albumin at least 3.0 mg/dL;
6. Provide tumor tissue, blood, and peritoneal lavage fluid samples;
7. Willing to accept long-term follow-up;
8. Ability to understand and sign a written informed consent before the trial procedure.

Exclusion Criteria

1. Currently participating in or receiving other clinical trial treatment;
2. Contraindications to investigational chemotherapy regimen including allergies to any of the chemotherapy medications;
3. Active infection requires systemic treatment;
4. Patients with poor compliance;
5. Patients who undergo non-curative surgery;
6. History of other malignant neoplasm within 5 years, except for early-stage skin cancer;
7. Pregnant or breast-feeding female;
8. Patients who have received neoadjuvant therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of peritoneal metastasis | Two years after surgery.
  The incidence of peritoneal metastasis.

SECONDARY OUTCOMES:
Peritoneal metastasis-free survival | Two years after surgery.
  The time from surgery to peritoneal metastasis.
Disease-free survival | Three years after surgery.
  The time from surgery to either recurrence or relapse of cancer, or death.
Overall survival | Three years after surgery.
  The time from surgery to death or the last follow-up date.
The safety | Ninety days after surgery.
  Adverse event and complications related to intraperitoneal chemotherapy. Adverse event is defined by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Complications will be recorded and graded according to the modified Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No